CLINICAL TRIAL: NCT04667104
Title: A Phase 2, Open-label, Single-arm, Multicenter Study to Assess Efficacy, Safety, Tolerability, and Pharmacokinetics of Treatment With JNJ-73763989, JNJ-56136379, Nucleos(t)Ide Analogs, and Pegylated Interferon Alpha-2a in Virologically Suppressed Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Study of JNJ-73763989, JNJ-56136379, Nucleos(t)Ide Analogs, and Pegylated Interferon Alpha-2a in Virologically Suppressed Participants With Chronic Hepatitis B Virus Infection
Acronym: PENGUIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108928; 2020-003956-34 (EudraCT Number); 73763989PAHPB2006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-12-09; First posted 2020-12-14 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; tenofovir alafenamide; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Period (TP) 1 (JNJ-73763989 + Nucleos(t)ide Analog)+ TP 2 (TP 1+PegIFN-alpha2a) (Experimental): Participants will receive combination treatment with JNJ-73763989+ nucleos(t)ide analog (NA) for 12 weeks during Treatment Period 1 and the participants who meet the eligibility criteria for PegIFN-alpha2a at Week 12 will receive combination treatment with JNJ-73763989 + NA plus PegIFN-α2a for 12 weeks during Treatment Period 2.
  Interventions: Drug: JNJ-73763989; Drug: Tenofovir disoproxil; Drug: Tenofovir alafenamide (TAF); Drug: Entecavir (ETV) monohydrate; Drug: PegIFN-alpha2a

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 injection will be administered subcutaneously once every 4 weeks.
  Other Names: JNJ-3989
Drug: Tenofovir disoproxil — Tenofovir disoproxil film-coated tablet will be administered orally once daily.
Drug: Tenofovir alafenamide (TAF) — TAF film-coated tablet will be administered orally once daily.
Drug: Entecavir (ETV) monohydrate — ETV monohydrate film-coated tablet will be administered orally once daily.
Drug: PegIFN-alpha2a — PegIFN-alpha2a injection will be administered subcutaneously once weekly.

SUMMARY:
The purpose of this study is to evaluate the efficacy in terms of hepatitis B surface antigen (HBsAg) levels of the study intervention (that is, JNJ-73763989 + JNJ-56136379 + nucleos[t]ide analog [NA] and pegylated interferon alpha-2a [PegIFN-alpha2a]).

DETAILED DESCRIPTION:
This study is an intervention specific appendix to the Hepatitis B wings platform trial (PLATFORMPAHPB2001). The study title reflects the original study design and JNJ-56136379 (JNJ-6379) was initially part of the study intervention but has been removed as part of amendment 3 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B virus (HBV) infection, hepatitis B e Antigen (HBeAg) positive or negative with suppressed viral replication under nucleos(t)ide analogue treatment for at least 6 months prior to screening
* Medically stable based on physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Body mass index (BMI) between 18.0 and 35.0 kilogram per meter square (kg/m^2), extremes included
* Must have serum HBsAg greater than (>) 100 international units per milliliter (IU/mL) at screening, as assessed by quantitative HBsAg assay
* Must have a fibroscan stiffness measurement less than or equal to (<=) 9.0 Kilopascal (kPa) at screening

Exclusion Criteria:

* Evidence of hepatitis A, C, D or E virus infection or human immunodeficiency, virus type 1 (HIV) or HIV-2 infection at screening
* History or evidence of clinical signs or symptoms of hepatic decompensation, including but not limited to: portal hypertension, ascites, hepatic encephalopathy, esophageal varices
* Evidence of liver disease of non-HBV etiology
* Participants with a history of malignancy within 5 years before screening
* Contraindications to the use of pegylated interferon alpha-2a

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- Japan (2):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Osaka University Hospital, Suita-shi
- New Zealand (2):
  - New Zealand Clinical Research, Auckland
  - Middlemore Clinical Trials, Papatoetoe
- Poland (4):
  - Neutrum Lekarze M.Hlebowicz i Partnerzy spolka partnerska, Gdansk
  - ID Clinic, Mysłowice
  - Wojewodzki Szpital Zakazny w Warszawie, Warsaw
  - Przychodnia EuroMediCare Wroclaw Lowiecka, Wroclaw
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Gane E, Janczewska E, Takehara T, Chuang WL, Peng CY, Hlebowicz M, Asahina Y, Chang TT, Kalmeijer R, Jezorwski J, Kim G, Anastasiou Z, Kakuda TN, Verbinnen T, Pehlivanov N, Bakala A, Lenz O, Biermer M. Peginterferon-alpha-2a add-on to treatment with siRNA JNJ-73763989 in virologically suppressed chronic hepatitis B: The phase II PENGUIN study. JHEP Rep. 2025 Jul 9;7(10):101516. doi: 10.1016/j.jhepr.2025.101516. eCollection 2025 Oct. PMID 40919077

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Week 12, participants were assessed for pegylated interferon alpha 2a (PegIFN-alpha2a) eligibility criteria and those who did not meet the criteria continued in Treatment Period 1 (TP 1) until Week 24 and those who met the criteria entered Treatment Period 2 (TP 2). After Week 12, one participant continued with TP1 regimen during TP2 until Week 24. As of Protocol Amendment 3, JNJ-56136379 was stopped immediately as study drug and study continued with JNJ-73763989, PegIFN alpha 2a & NA only.
Groups:
- TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA: Participants received a single dose of JNJ-73763989 (JNJ-3989) 200 milligrams (mg) as a subcutaneous injection (SC) every 4 weeks (Q4W) along with JNJ-56136379 (JNJ-6379) 250 mg tablet once daily (QD) and nucleos(t)ide analog (NA) treatment (either entecavir[ETV] 0.5 mg, tenofovir disoproxil fumarate[TDF] 245 mg, or tenofovir alafenamide[TAF] 25 mg) QD up to 12 weeks in TP 1. Participants enrolled until Protocol Amendment 3, also received single dose of JNJ-56136379 250 mg orally as part of their study intervention. Participants enrolled after protocol amendment 3, received JNJ-3989 + PegIFN-alpha 2a + NA only. Participants were assessed for eligibility criteria for PegIFN-alpha 2a at Week 12. Participants who met the criteria entered TP 2.
- TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA: Participants who met the eligibility criteria for PegIFN-alpha2a (Participants who did not have disorders including but not limited to: autoimmune disorders, bone marrow suppression, hypoglycemia, hyperglycemia, diabetes mellitus) at Week 12 received combination treatment with JNJ-73763989 200 mg SC injection Q4W along with NA treatment (either ETV 0.5 mg, TDF 245 mg, or TAF 25 mg) QD up to Week 24 plus PegIFN-alpha 2a 180 micrograms (mcg) once weekly (QIW) during TP 2. Participants enrolled until Protocol Amendment 3, also received single dose of JNJ-56136379 250 mg orally as part of their study intervention. Participants enrolled after Protocol Amendment 3, received JNJ-73763989 + PegIFN alpha 2a + NA only.
- Follow-Up (FU) Period-nucleos(t)Ide Analog (NA): At Week 24, prior to follow-up period, all participants stopped treatment with JNJ-73763989 + JNJ-56136379 + PegIFN-alpha2a. Participants who met the protocol-defined NA treatment completion criteria (hepatitis B surface antigen [HBsAg] <10 international units/millilitre [IU/mL], and hepatitis B e antigen [HBeAg]-negative, and hepatitis B virus deoxyribonucleic acid [HBV DNA] <20 IU/mL <lower limit of quantification [LLOQ], and alanine aminotransferase [ALT] <3*Upper limit of normal [ULN]) at Week 24, stopped NA at Week 26 (that is follow up Week 2). Participants who did not meet NA completion criteria continued NA treatment during the follow-up period up to follow-up Week 48 (with window period of +/- 4 days that is up to Week 72.4).
Period: TP 1: From Week 1 to Week 12
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Started | 48 | 0 | 0
Completed | 48 | 0 | 0
Not Completed | 0 | 0 | 0
Period: TP 2: From Week 12 to Week 24
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Started | 0 | 48 | 0
Completed | 0 | 48 | 0
Not Completed | 0 | 0 | 0
Period: FU:Week 24 to FU Week 48 (i.e.Week 72.4)
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Started | 0 | 0 | 48
Completed | 0 | 0 | 47
Not Completed | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (1.47) [lower limit 1.47]
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 48
  From 65 to 84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 34
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Reduction of at Least 2 log10 International Unit/Millilitres (IU/mL) in Hepatitis B Surface Antigen (HBsAg) Levels From Baseline to Week 24
Description: Percentage of participants with a reduction of at least 2 log10IU/mL in HBsAg levels from baseline to Week 24 were reported. A responder was defined as a participant with reduction of at least 2 log10 IU/mL in HBsAg levels from baseline at Week 24.
Time Frame: From Baseline (Day 1) to Week 24
Population: Full Analysis Set (FAS) included all participants who were enrolled and who received at least 1 dose of study intervention within this intervention-specific appendix (ISA). Data for this outcome measure was planned to be collected and analyzed for specified arm only.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA
Number analyzed (Participants) | 48
percentage of participants | 64.6 (51.73) [51.73 to 76.02]

2. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability
Description: Percentage of participants with TEAEs were reported. An adverse event (AE) was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs were AEs with onset during the intervention period or follow-up period or that were a consequence of a pre-existing condition that had worsened since baseline.
Time Frame: Treatment Period 1: From Baseline (Day 1) up to Week 12; Treatment Period 2: From Week 12 up to Week 24; Follow-Up Period: From Week 24 up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
percentage of participants | 52.1 | 87.5 | 60.4

3. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs were AEs with onset during the intervention period or follow-up period or that were a consequence of a pre-existing condition that had worsened since baseline. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
percentage of participants | 0 | 2.1 | 8.3

4. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs as a Measure of Safety and Tolerability
Description: Number of participants with clinically significant abnormalities in vital signs (pulse rate, and blood pressure [systolic and diastolic]) were reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Findings as a Measure of Safety and Tolerability
Description: Number of participants with clinically significant abnormalities in laboratory findings (including hematology, blood biochemistry, and urinalysis) were reported. Only parameters in which any participant had abnormality are reported below.
Time Frame: as for outcome 2
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this endpoint and "n"(number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
Participants
  Treatment-emergent (TE)-Grade 3 ALT elevations | 1 | 1 | 1
  TE-Grade 3 total bilirubin elevations | 0 | 0 | 1
  TE-Grade 3 direct bilirubin elevations | 0 | 0 | 2
  Treatment-emergent-High serum indirect bilirubin | 0 | 0 | 3
  Renal complications-eGFR Decreases | 0 | 0 | 0
  Hematology-low absolute neutrophil count Grade 1 | 1 | 13 | 2
  Hematology-low absolute neutrophil count Grade 2 | 0 | 2 | 1
  Hematology-low absolute neutrophil count Grade 3 | 0 | 3 | 0
  Hematology-low absolute neutrophil count Grade 4 | 0 | 1 | 0
  Hematology-low absolute lymphocyte count Grade 1 | 1 | 1 | 0
  Hematology-low absolute lymphocyte count Grade 2 | 1 | 3 | 0
  Hematology-low absolute lymphocyte count Grade 3 | 0 | 3 | 2
  Hematology-low absolute lymphocyte count Grade 4 | 0 | 1 | 1
  Hematology-decreased platelets of Grade 1 | 0 | 20 | 8
  Hematology-decreased platelets of Grade 2 | 0 | 5 | 0
  Hematology-low hemoglobin Grade 2 | 0 | 0 | 1
  Hematology-low WBC count of Grade 1 | 0 | 14 | 5
  Hematology-low WBC count of Grade 2 | 0 | 6 | 1
  Hematology-low WBC count of Grade 3 | 0 | 2 | 0
  Chemistry-LDL cholesterol Grade 3 | 2 | 1 | 2
  Chemistry-eGFR creatinine low Grade 3 elevation | 1 | 0 | 0
  Chemistry-eGFR Cystatin C low Grade 3 elevation | 0 | 1 | 2
  Chemistry-Grade 3 elevations in triglycerides | 0 | 2 | 0
  Chemistry-Grade 3 elevation amylase | 0 | 0 | 1
  Chemistry-Grade 3 elevation direct bilirubin high | 0 | 0 | 2
  Chemistry-lipaseGrade 4 elevation | 0 | 0 | 1
  Urinalysis-Grade 1 glycosuria | 0 | 0 | 1
  Urinalysis-Grade 1 hematuria | 0 | 1 | 1
  Urinalysis-Grade 2 hematuria | 1 | 1 | 1
  Urinalysis-Grade 1 proteinuria | 2 | 5 | 4
  Urinalysis-Grade 2 proteinuria | 1 | 1 | 1

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECGs) as a Measure of Safety and Tolerability
Description: Number of participants with clinically significant abnormalities in 12- lead ECGs (heart rate, PR, QRS and QT corrected [QTc]) were reported.
Time Frame: Treatment Period 1: From Baseline (Day 1) up to Week 12; Treatment Period 2: From Week 12 up to Week 24; Follow-Up Period: From Week 24 up to Week 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination as a Measure of Safety and Tolerability
Description: Number of participants with clinically significant abnormalities in physical examination were reported.
Time Frame: Treatment Period 1: From Baseline (Day 1) up to Week 12; Treatment Period 2: From Week 12 up to Week 24
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received. Data for this outcome measure was not planned to be collected and analyzed for Follow-Up Period as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA
Number analyzed (Participants) | 48 | 48
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormalities in Ophthalmic Examination as a Measure of Safety and Tolerability
Description: Number of participants with abnormalities in Ophthalmic examination were planned to be reported.
Time Frame: Treatment Period 1: From Baseline (Day 1) up to Week 12; Treatment Period 2: From Week 12 up to Week 24
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received. Data for this outcome measure was planned to be collected and analyzed at TP 1 and TP 2 for participants with diabetes/hypertension only. Since no subject had diabetes/hypertension hence data for this OM was not collected and analyzed as pre-specified in protocol.
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants Meeting the Protocol-defined Nucleos(t)Ide Analog (NA) Treatment Completion Criteria at End of Study Intervention (EOSI)
Description: Percentage of participants meeting the protocol-defined NA treatment completion criteria at EOSI were reported. NA treatment completion criteria are defined based on laboratory results at Week 24 were; HBsAg <10 IU/mL; HBeAg-negative; HBV DNA <20 IU/mL, that is, lower limit of quantification(LLOQ); alanine aminotransferase(ALT) <3*ULN.
Time Frame: At Week 24 (EOSI)
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA. Data for this outcome measure was not planned to be collected and analyzed for Treatment Period 1 and Follow-Up period as pre-specified in protocol.
Measure: Number; unit: percentage of participants
Arm/Group | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA
Number analyzed (Participants) | 48
percentage of participants | 31.3

10. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Levels Below Different Cut-offs
Description: Percentage of participants with HBeAg levels below different cut-offs were reported. The cut-offs for HBeAg levels were as followed:< 100 IU/mL, < 10 IU/mL, < 1 IU/mL, < LLOQ (0.11 IU/mL).
Time Frame: as for outcome 2
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 11 | 11 | 11
percentage of participants
  < LLOQ (0.11 IU/mL) | 36.4 | 27.3 | 27.3
  < 1 IU/mL | 90.9 | 100.0 | 81.8
  < 10 IU/mL | 100.0 | 100.0 | 100.0
  < 100 IU/mL | 100.0 | 100.0 | 100.0

11. Secondary Outcome: Percentage of Participants With HBsAg Levels Below Different Cut-offs
Description: Percentage of participants with HBsAg levels below different cut-offs were reported. The cut-offs for HBsAg level were: <1000 IU/mL, <100 IU/mL, <10 IU/mL, <1 IU/mL, <LLOQ (0.05 IU/mL).
Time Frame: as for outcome 2
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA.
Measure: Number; unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
percentage of participants
  <LLOQ (0.05 IU/mL) | 0 | 2.1 | 2.1
  <1 IU/mL | 4.2 | 6.3 | 2.1
  <10 IU/mL | 12.5 | 47.9 | 4.2
  <100 IU/mL | 58.3 | 91.7 | 27.1
  <1000 IU/mL | 89.6 | 97.9 | 68.8

12. Secondary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Levels Below Different Cut-offs
Description: Percentage of participants with HBV DNA levels below cut-offs were reported. The cut-offs for HBV DNA were as follows: <LLOQ (=20 IU/mL) target detected or not detected, < LLOQ target not detected, and < LLOQ target detected, <60 IU/mL, <100 IU/mL, <200 IU/mL, <1000 IU/mL, <2000 IU/mL, <20000 IU/mL.
Time Frame: as for outcome 2
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA.
Measure: Number; unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
percentage of participants
  < LLOQ for target detected and not detected | 95.8 | 75.0 | 81.3
  < LLOQ for target not detected | 52.1 | 27.1 | 54.2
  < LLOQ for target detected | 43.8 | 47.9 | 27.1
  < 60 IU/mL | 100.0 | 89.6 | 83.3
  < 100 IU/mL | 100.0 | 95.8 | 83.3
  < 200 IU/mL | 100.0 | 97.9 | 85.4
  < 1000 IU/mL | 100.0 | 100.0 | 89.6
  < 2000 IU/mL | 100.0 | 100.0 | 93.8
  < 20000 IU/mL | 100.0 | 100.0 | 97.9

13. Secondary Outcome: Percentage of Participants With ALT Levels Greater Than or Equal to (>=) 3*ULN
Description: Percentage of participants with ALT levels below >=3*ULN cut-off were reported.
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 3 | 3 | 3
percentage of participants | 33.3 | 33.3 | 66.7

14. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion
Description: Percentage of participants with HBeAg seroconversion were reported. Seroconversion of HBeAg is defined as having achieved HBeAg seroclearance (as HBeAg level <LLOQ [0.11 IU/mL]) and appearance of anti-HBe antibodies, defined as baseline anti-HBe antibodies with a negative result and a post-baseline assessment with positive result.
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 11 | 11 | 11
percentage of participants | 0 | 10.0 | 20.0

15. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion
Description: Percentage of participants with HBsAg seroconversion were reported. Seroconversion of HBsAg was defined as having achieved HBsAg seroclearance (defined as HBsAg <LLOQ [0.05 IU/mL]) and appearance of anti-HBs antibodies.
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 45 | 46 | 46
percentage of participants | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline Over Time in HBsAg Levels
Description: Change from baseline over time in HBsAg levels were reported. The baseline assessment was defined as the last observed non-missing measurement before the date and time of the first administration of any of study agent.
Time Frame: Treatment Period 1: From Baseline (Day 1) up to Week 12; Treatment Period 2: From Baseline (Day 1) up to Week 24; Follow-Up: From Baseline (Day 1) up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4)
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA.
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
log10 IU/mL | -1.43 (0.070) [lower limit 0.070] | -2.18 (0.084) [lower limit 0.084] | -0.71 (0.092) [lower limit 0.092]

17. Secondary Outcome: Change From Baseline Over Time in HBeAg Levels
Description: Change from baseline over time in HBeAg levels were reported. The baseline assessment was defined as the last observed non-missing measurement before the date and time of the first administration of any of study agent.
Time Frame: as for outcome 16
Population: as for outcome 10
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 11 | 11 | 11
log10 IU/mL | -0.68 (0.087) [lower limit 0.087] | -0.72 (0.106) [lower limit 0.106] | -0.53 (0.112) [lower limit 0.112]

18. Secondary Outcome: Change From Baseline Over Time in HBV DNA Levels
Description: Change from baseline over time in HBV DNA levels were reported. The baseline assessment was defined as the last observed non-missing measurement before the date and time of the first administration of any of study agent.
Time Frame: as for outcome 16
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA.
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
log10 IU/mL | 0.03 (0.032) | 0.28 (0.059) | 0.36 (0.145)

19. Secondary Outcome: Time to First Occurrence of HBsAg Seroclearance
Description: Time to first occurrence of HBsAg seroclearance were reported in median time. Time to first occurrence of the HBsAg seroclearance was defined as the number of days between the date of first study intervention intake and the date of first occurrence of the HBsAg seroclearance.
Time Frame: From Baseline (Day 1) up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4)
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA. Data for this endpoint was planned to be collected and analyzed in a single arm.
Measure: Median (Full Range); unit: weeks
Groups:
- Pooled (JNJ-3989 200mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA): Participants received JNJ-3989 200 mg as SC Q4W along with JNJ-6379 250 mg tablet QD and NA treatment (either ETV 0.5 mg, TDF 245 mg, or TAF 25 mg QD up to 12 weeks in TP1. At Week 12, participants who met eligibility criteria for PegIFN-alpha 2a entered TP2. Participants in TP2 received combination treatment of JNJ-3989 200 mg SC injection Q4W with NA treatment up to Week 24 plus PegIFN-alpha 2a 180 mcg Q1W. At Week 24, before follow-up period, participants stopped JNJ-3989 + JNJ-6379 + PegIFN-alpha2a. At Week 26, those who met the NA treatment completion criteria stopped NA (follow up Week 2) and those who did not meet criteria continued NA treatment in follow-up period up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4). Participants enrolled until Protocol Amendment 3 (PA3), also received JNJ-6379 250 mg orally as intervention in TP1 and TP2 and those enrolled after PA3, received only JNJ-3989 + PegIFN alpha 2a + NA during study.
Arm/Group | Pooled (JNJ-3989 200mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA)
Number analyzed (Participants) | 48
weeks | NA [NA to NA] — NA indicates that median [range] data were not estimable as at least 50% participants did not reach HBsAg seroclearance.

20. Secondary Outcome: Time to First Occurrence of HBeAg Seroclearance
Description: Time to first occurrence of HBeAg seroclearance were reported in median time. Time to first occurrence of the HBeAg seroclearance is defined as the number of days between the date of first study intervention intake and the date of the first occurrence of the HBeAg seroclearance.
Time Frame: From Baseline (Day 1) up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4)
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA. Here "N" (number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed in a single arm.
Measure: Median (Full Range); unit: weeks
Arm/Group | Pooled (JNJ-3989 200mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA)
Number analyzed (Participants) | 11
weeks | 14.1 [4.1 to 72.4]

21. Secondary Outcome: Time to First Occurrence of HBV DNA < LLOQ
Description: Time to first occurrence of HBV DNA < LLOQ (20 IU/mL) were reported in median time. Time to first occurrence of the HBV DNA < LLOQ is defined as the number of days between the date of first study intervention intake and the date of the first occurrence of the HBV DNA < LLOQ.
Time Frame: From Baseline (Day 1) up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4)
Population: as for outcome 19
Measure: Median (Full Range); unit: weeks
Arm/Group | Pooled (JNJ-3989 200mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA)
Number analyzed (Participants) | 48
weeks | 4.1 [2.9 to 32.3]

22. Secondary Outcome: Percentage of Participants With Virologic Breakthrough
Description: Percentage of Participants with virologic breakthrough were reported. It was defined as confirmed on-treatment (the time period during which the participant received any of the study treatments) HBV DNA increase by >1 log10 IU/mL from nadir or confirmed on-treatment HBV DNA level >200 IU/mL in participants who had HBV DNA level <LLOQ (20 IU/mL) of the HBV DNA assay. Confirmed means that the criteria were fulfilled at 2 or more consecutive time points or at the last observed time point.
Time Frame: Treatment Period 1: From Baseline (Day 1) up to Week 12; Treatment Period 2: From Week 12 up to Week 24; Follow-Up: From Week 24 up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 38
percentage of participants | 0 | 0 | 0

23. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance at Week 48 Without Re-starting NA Treatment
Description: Percentage of participants with HBsAg seroclearance at Week 48 (i.e., 24 weeks after completion of all study interventions at Week 24) without re-starting NA treatment were reported. HBsAg seroclearance was defined as [quantitative] HBsAg <LLOQ (0.05 IU/mL).
Time Frame: At Week 48 (24 weeks after completion of all study interventions at Week 24)
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA. Data for this outcome measure was planned to be collected and analyzed for Follow-Up Period only as pre-specified in protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48
percentage of participants | 0

24. Secondary Outcome: Percentage of Participants With HBV DNA < LLOQ at Week 48 Without Re-starting NA Treatment
Description: Percentage of participants with HBV DNA <LLOQ (20 IU/mL) at Week 48 (that is, 24 weeks after completion of all study interventions at Week 24) without re-starting NA treatment were reported.
Time Frame: At Week 48 (24 weeks after completion of all study interventions at Week 24)
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for Follow-Up Period only as pre specified in protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 10
percentage of participants | 30.0

25. Secondary Outcome: Percentage of Participants With Biochemical Flares
Description: Percentage of participants with biochemical flares were reported. On-treatment biochemical flare was defined as confirmed ALT and/or AST >=3*ULN and >=3*nadir, while the participant received any of the study interventions. Off-treatment biochemical flare was defined as confirmed ALT and/or AST =3*ULN and =3*nadir, while the participants did not receive any of the study interventions (Off treatment, including NA).
Time Frame: as for outcome 22
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure and "n"(number analyzed) signifies number of participants analyzed at specified categories. No participant was available for the analysis where "n=0".
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 48 | 48 | 48
percentage of participants
  On-Treatment: number analyzed (Participants) | 48 | 48 | 38
  On-Treatment | 0 [0 to 6.05] | 4.2 [0.75 to 12.54] | 0 [0 to 7.58]
  Off-Treatment: number analyzed (Participants) | 0 | 0 | 15
  Off-Treatment |  |  | 0 [0 to 0]

26. Secondary Outcome: Percentage of Participants With Virologic Flares
Description: Percentage of participants with virologic flares were reported. Virologic flare was defined as confirmed HBV DNA >peak threshold (lowest peak to qualify as virologic flare was HBV DNA >200 IU/mL) in participants who were off-treatment. Off-treatment was defined as the time period after stopping all study treatments (including NA) and had HBV DNA <LLOQ (20 IU/mL) at the last observed time point on all study interventions.
Time Frame: Follow-Up Period: From Week 24 up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4)
Population: FAS included all participants who were enrolled and who received at least 1 dose of study intervention within this ISA. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for Follow-Up period only as pre-specified in protocol.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 15
percentage of participants | 33.3 (14.17) [14.17 to 57.74]

27. Secondary Outcome: Number of Participants Requiring NA Re-treatment
Description: Number of participants requiring NA re-treatment based on failure in NA treatment completion criteria (HBsAg <10 IU/mL, and HBeAg-negative, and HBV DNA < LLOQ (20 IU/mL), and ALT <3*ULN) were reported.
Time Frame: Follow-Up Period: From Week 24 up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 15
Participants | 4

28. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of JNJ-73763989 (JNJ-73763976 and JNJ-73763924)
Description: The maximum observed plasma concentrations (Cmax) of JNJ-73763989 (JNJ-73763976 and JNJ-73763924) were reported.
Time Frame: Treatment Period 1: Day 1 Week 1; Treatment Period 2: Day 1, Week 12
Population: Pharmacokinetics(PK) analysis set included participants who received at least 1 dose of study intervention and had at least 1 valid blood sample drawn for PK analysis. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for TP1 and TP2 only as specified in protocol.
Measure: Mean (Standard Deviation); unit: nanograms/milliliters (ng/mL)
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA
Number analyzed (Participants) | 5 | 5
nanograms/milliliters (ng/mL)
  JNJ-73763976 | 1338 (971) | 928 (692)
  JNJ-73763924 | 271 (197) | 185 (130)

29. Secondary Outcome: Plasma Concentration 24 Hours After Administration (C24h) of JNJ-73763989 (JNJ-73763976 and JNJ-73763924)
Description: Plasma concentration 24 hours (C24h) after administration of JNJ-73763989 (JNJ-73763976 and JNJ-73763924) were reported.
Time Frame: Treatment Period 1: Day 1 Week 1; Treatment Period 2: Day 1, Week 12
Population: PK Analysis Set included all participants who received at least 1 dose of study intervention and had at least 1 valid blood sample drawn for PK analysis. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for TP 1 and TP 2 as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA
Number analyzed (Participants) | 5 | 5
ng/mL
  JNJ-73763976 | 309 (145) | 390 (162)
  JNJ-73763924 | 38.7 (16.2) | 57.4 (15.9)

30. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-73763989 (JNJ-73763976 and JNJ-73763924)
Description: Time to reach maximum observed plasma concentration (Cmax) (Tmax) of JNJ-73763989 (JNJ-73763976 and JNJ-73763924) were reported.
Time Frame: Treatment Period 1: Day 1, Week 1; Treatment Period 2: Day 1, Week 12
Population: PK analysis set included all participants who received at least 1 dose of study intervention and had at least 1 valid blood sample drawn for PK analysis. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for TP1 and TP2 as pre-specified in protocol.
Measure: Median (Full Range); unit: hours
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA
Number analyzed (Participants) | 5 | 5
hours
  JNJ-73763976 | 5.50 [2.00 to 6.20] | 6.00 [2.00 to 23.58]
  JNJ-73763924 | 2.00 [1.00 to 6.00] | 4.02 [0.50 to 7.72]

31. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hour (AUC[0-24]h) of JNJ-73763989 (JNJ-73763976 and JNJ-73763924)
Description: Area under the plasma concentration versus time curve from time 0 to 24 hours (AUC[0-24]h) of JNJ-73763989 (JNJ-73763976 and JNJ-73763924) were reported.
Time Frame: Treatment Period 1: Day 1, Week 1; Treatment Period 2: Day 1, Week 12
Population: PK analysis set: participants who received at least 1 dose of study intervention and had at least 1 valid blood sample drawn for PK analysis. Here "N" (number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for TP1 and TP2 as specified in protocol.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA
Number analyzed (Participants) | 5 | 5
ng*h/mL
  JNJ-73763976 | 18635 (10983) | 13580 (8598)
  JNJ-73763924 | 3342 (1919) | 2466 (1432)

ADVERSE EVENTS:
Time Frame: Treatment Period 1: From Baseline (Day 1) up to Week 12; Treatment Period 2: From Week 12 up to Week 24; Follow-Up: From Week 24 up to follow-up Week 48 (with window period of +/- 4 days, that is Week 72.4)
Description: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Arm/Group | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/48 | 4/48
Other Adverse Events (participants affected / at risk) | 12/48 | 35/48 | 20/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA (N=48) | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA (N=48) | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA) (N=48)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic Mass (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TP 1:JNJ-73763989 200 mg+JNJ-56136379 250 mg+NA (N=48) | TP 2:JNJ-3989 200 mg+JNJ-6379 250 mg+PegIFN-alpha2a 180 mcg+NA (N=48) | Follow-Up (FU) Period-nucleos(t)Ide Analog (NA) (N=48)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (6) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (3) | 5 (5) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 6 (7) | 0 (0)
Injection Site Erythema (General disorders) | 1 (1) | 7 (10) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 15 (18) | 2 (2)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 13 (13)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (7)
Alanine Aminotransferase Increased (Investigations) | 1 (2) | 3 (4) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 4 (7) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (9) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04667104/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT04667104/SAP_001.pdf